CLINICAL TRIAL: NCT06545227
Title: An Observational Nested Multicenter Cohort Study of Early Versus Late Monitoring Among Pregnant Women With a History of Gestational Diabetes
Brief Title: Early Versus Late Monitoring Among Pregnant Women With a History of Gestational Diabetes
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Bold insight (Unknown); DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 304605
Record Dates: First submitted 2024-02-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Complications; Gestational Diabetes
MeSH Terms: conditions — Pregnancy Complications; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early monitoring group: Women who are testing blood glucose four times a day from 28 weeks.
  Interventions: Other: Collection of urine, maternal blood at baseline and 28 weeks in a subset of women (n=25); Other: Collection of umbilical cord blood, placental samples and cord tissue in a subset of women (n=25); Other: Maternal and neonatal outcome data collection for all women in the study
- Late monitoring group: Women who have an oral glucose tolerance test at 28-32 weeks.
  Interventions: Device: continuous blood glucose monitoring in a subset of women (n=25) in the early monitoring group.; Other: Collection of urine, maternal blood at baseline and 28 weeks in a subset of women (n=25); Other: Collection of umbilical cord blood, placental samples and cord tissue in a subset of women (n=25); Other: Maternal and neonatal outcome data collection for all women in the study

INTERVENTIONS:
Device: continuous blood glucose monitoring in a subset of women (n=25) in the early monitoring group. — To continuously monitor blood glucose from baseline to 28 weeks to determine if if there is hyperglycaemia in a subset of women (n=25)
  Groups: Late monitoring group
Other: Collection of urine, maternal blood at baseline and 28 weeks in a subset of women (n=25) — To study maternal metabolome
Other: Collection of umbilical cord blood, placental samples and cord tissue in a subset of women (n=25) — To study mesenchymal stem cell differentiation, change in fetal epigenetic and placental signalling pathways.
Other: Maternal and neonatal outcome data collection for all women in the study — Data for maternal and neonatal outcomes will be collected

SUMMARY:
The goal of this study investigate if pregnant women with a history of gestational diabetes (GDM) have better pregnancy outcomes if they test their blood glucose four times a day early in the pregnancy versus having an oral glucose tolerance test later in the pregnancy at 28 weeks in their current pregnancy.

Population being studied:

All pregnant women who had a history of GDM in a previous pregnancy

Study groups:

1. Women who are being managed in the pregnancy with early blood glucose monitoring (early monitoring group)
2. Women who are being managed with an oral glucose tolerance test at 28-32 weeks (late monitoring group)

This study has two parts (i) observational and (ii) mechanistic or laboratory based.

In the observational part of the study, data will be collected as standard of care across different obstetric units and this data will be used to:

1. compare the outcomes of the women such as need for labour to be induced, caesarean section rates, blood loss, need for treatment of their blood glucose with metformin or insulin, HbA1c values
2. compare the outcomes of the offspring such as birth weight centiles, shoulder dystocia or birth trauma, hypoglycaemia, jaundice and if admitted to the neonatal unit.

The mechanistic or laboratory part of the study is aimed at studying how the two different treatment approaches affect:

1. the metabolome of the pregnant woman - urine and blood samples collected at two time points will be used and mass spectrometry used to determine the amino acid and lipid profiles.
2. the microbiome differs between both groups
3. the pathways that regulate insulin in the placenta
4. the ability of the cells in the umbilical cord differentiate into the different fat cells.

DETAILED DESCRIPTION:
Gestational diabetes rates are globally increasing and it is now well known that women who had gestational diabetes have a recurrent risk ranging from 35.5% to 70% in a future pregnancy. Some of these women may have preexisting type 2 diabetes or glucose intolerance There is also now convincing evidence that the women with GDM are at increased risk of T2DM and cardiovascular disorders. GDM can also affect the health of the offspring and associated with an increased risk of future obesity, diabetes and cardiovascular disorders, possibly modulated through altered epigenetics of the fetus. The recent NICE guidance has recommended that women with a history of GDM should be offered early pregnancy glucose monitoring or testing with oral glucose tolerance test at 24-28 weeks. Gestational diabetes is associated with derangement in amino acid and lipid pathways and these changes can be demonstrated several weeks prior to the diagnosis of GDM. Similarly, both candidate gene and genome wide studies have reported that GDM exposure is associated with significant changes in the infant's or child's DNA methylation, with a recent meta-analysis of seven pregnancy cohorts identified differentially methylated regions (DMRs) associated with GDM within OR2L13 and CYP2E1. Others have also been able to demonstrate that GDM-associated methylation is associated with offspring obesity and T2DM.

There is emerging evidence that in pregnancy gestational diabetes can occur as early as the first trimester. However in clinical practice, screening and diagnosis does not occur until 28 weeks in the pregnancy, suggesting that in some cases the fetus may be exposed to undetected hyperglycaemia much earlier. There is varying practice in how a pregnant women with a history of GDM is managed in a future pregnancy. Some are offered early capillary blood glucose testing four times a day as early as 10 weeks (early monitoring), while others are offered diagnostic testing with an oral glucose tolerance test at 28 weeks (late monitoring). This study was designed to compare the pregnancy outcomes between the early and the late monitoring approaches to determine which is more effective in modulating the maternal metabolome, placental insulin signalling pathways and offspring DNA methylation. Equally important the multi-centre observational arm will allow comparison of maternal and neonatal outcomes between both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age >16
2. Pregnant
3. Previous pregnancy with gestational diabetes diagnosed by an Oral Glucose Tolerance Test
4. Singleton pregnancy

Exclusion Criteria:

Women with the following risk factors will be excluded:

1. Multiple pregnancy
2. History of bariatric surgery
3. Taking metformin or other oral hypoglycaemic agents
4. HbA1c more than or equal to 48

Ages: 17 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — pregnant women
Study Population: All pregnant women with a history of gestational diabetes in a previous pregnancy diagnosed by an oral glucose tolerance test.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the maternal metabolome between the early monitoring group and the late monitoring group. | 12 months
  Mass spectrometry will be used to study and analyse roughly 200 aqueous metabolites from glycolysis, TCA cycle, amino acid metabolism, nucleotides, beta-oxidation and the pentose phosphate pathway, with quantification against stable isotope labelled standards
Comparison of the cord blood DNA methylation between the early monitoring group and the late monitoring group | 12 months
  Cord blood DNA methylation will be assessed using the Methylation EPIC BeadArray (850,000 CpG sites). We will identify DMCpGs and DMRs, together with the networks and transcriptional hubs associated with GDM and the potential mediators and pathways.

SECONDARY OUTCOMES:
Comparison of Maternal HbA1c in first and third trimesters | 12 months
  Data from clinical records will be used to compare between the two groups (i) HbA1c in first and third trimesters
Comparison of type of labour between both study groups | 12 months
  We will compared between both groups the rate of spontaneous labour, induced labours or caesarean section
Comparison of requirement for drug treatment with metformin or insulin between both groups | 12 months
  Clinical data on treatment with insulin and/or metformin will be recorded for both cohorts and compared
Comparison of rates of postpartum haemorrhage (>500mls blood) and third degree tears among both groups | 12 months
  Complications such as haemorrhage, and perineal trauma will be compared between groups
Comparison of the composite neonatal outcome between both groups | 12 months
  Data from clinical records will be used to record and compare the composite neonatal outcome (stillbirth, hypoglycaemia, jaundice, admission to neonatal unit)
Comparison of rates of shoulder dystocia between both study cohorts | 12 months
  Data on the number of cases of shoulder dystocia will be compared between the both study groups

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Singh, MBBS FRCOG, Study Chair — Imperial College London
Locations (1):
- Chelsea and Westminster Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared but anonymised and via peer review publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after study completed and will remain available for 12 months after
Access Criteria: Researchers undertaking similar research will be able to have access to the data and study documents.
  The data will be shared via email and will by anonymised The Chief investigator will review the request